CLINICAL TRIAL: NCT00552162
Title: NOTES Transvaginal Cholecystectomy and Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOTES HMO-CTIL; 21-2.11.07
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2016-04

CONDITIONS: Gallbladder Diseases; Appendicitis
MeSH Terms: conditions — Gallbladder Diseases; Appendicitis

ARMS (2):
- 1 (Active Comparator): NOTES Transvaginal cholecystectomy The gallbladder will be dissected free and will be removed through an incision in the vagina.
  Interventions: Procedure: NOTES Transvaginal Cholecystectomy
- 2 (Active Comparator): NOTES Transvaginal Appendectomy. The appendix will be dissected free and will be removed through an incision in the vagina.
  Interventions: Procedure: NOTES Transvaginal Appendectomy

INTERVENTIONS:
Procedure: NOTES Transvaginal Cholecystectomy — The gallbladder will be dissected free and will be removed through an incision in the vagina.
  Arms: 1
Procedure: NOTES Transvaginal Appendectomy — The appendix will be dissected free and will be removed through an incision in the vagina.
  Arms: 2

SUMMARY:
Natural Orifice Translumenal Endoscopic Surgery (NOTES) is considered by many leading expert surgeons to be the next step in MIS (Minimally Invasive Surgery). This is a rapidly evolving area of preclinical research and several groups worldwide are developing this surgical approach together with industry support. In this new surgical technique, abdominal operations are performed using the oropharynx, rectum, or vagina as the ports of entry to the peritoneal cavity instead of incisions on the abdominal wall. NOTES offers all the advantages of minimally invasive surgery (MIS) and also completely eliminates trauma to the abdominal wall and the numerous complications of abdominal wall incisions. A NOTES procedure eliminates any visible scar and could also potentially reduce post operative pain due to the elimination of abdominal wall trauma.

In this trial we intend to operate healthy women who need to undergo cholecystectomy or appendectomy. The operations will be performed through the vagina as the access port to the peritoneum and it will be monitored with laparoscopic vision for safety reasons.

ELIGIBILITY:
Inclusion Criteria for group #1 Transvaginal cholecystectomy:

1. Females between the ages of 18 and 50
2. Diagnosis of gallstone disease which requires cholecystectomy
3. ASA class 1

Exclusion Criteria for group #1 Transvaginal cholecystectomy:

1. Pregnant women
2. Morbidly obese patients (BMI > 35)
3. Patients who are taking immunosuppressive medications and/or immunocompromised
4. Patients with severe medical comorbidities will be excluded.
5. Patients with a presumed gallbladder polyps, mass or tumor
6. Patients with a history of prior open abdominal or transvaginal surgery.
7. Patients with a prior history of peritoneal or vaginal trauma
8. Patients with a history of ectopic pregnancy, pelvic inflammatory disease, or severe endometriosis
9. Patients with known common bile duct stones
10. Patients on blood thinners or aspirin or abnormal blood coagulation tests

Inclusion Criteria for group #2 Transvaginal appendectomy:

1. Clinical diagnosis of appendicitis
2. Emergency room evaluation within 36 hours of the onset of pain
3. ASA Classification

Exclusion Criteria for group #2 Transvaginal appendectomy:

1. pregnant women
2. Morbidly obese patients (BMI >35)
3. Patients who are taking immunosuppressive medications or are immunocompromised
4. Patients with evidence of an abdominal abscess or mass
5. Patients who present with a clinical diagnosis of sepsis or peritonitis
6. Patients who have a history of prior open abdominal surgery or prior transvaginal surgery.
7. Patients who endorse a history of ectopic pregnancy, pelvic inflammatory disease (PID), or severe endometriosis
8. Patients with diffuse peritonitis on clinical exam
9. Previous trauma to the perineal area
10. Patients on blood thinners or aspirin or abnormal blood coagulation tests

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06; Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
TO ASSESS THE SAFETY AND EFFICACY OF A NOVEL APPROACH TO MINIMALLY INVASIVE SURGICAL TECHNIQUES | continuous

SECONDARY OUTCOMES:
TO ASSESS PAIN ASSOCIATED WITH TRANSVAGINAL APPROACH | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Mintz, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Hadassah Medical Organization, Jerusalem